CLINICAL TRIAL: NCT03585114
Title: Prostate Cancer Monitoring Using [18F]DCFPyL and Blood Based Biomarkers
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Matthew Dallos, Assistant Professor of Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAR6032
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Intervention Model Description: Fifteen men will be recruited from Columbia University Medical Center.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PyL-PET (Experimental): Male participants diagnosed with metastatic castrate resistant prostate cancer (mCRPC) and are scheduled to start a new treatment will receive [F-18] DCFPyL PET/CT imaging before starting new treatment and after 6 weeks on treatment.
  Interventions: Drug: [F-18] DCFPyL; Procedure: PET/CT imaging

INTERVENTIONS:
Drug: [F-18] DCFPyL — [18F]DCFPyL will be used for study imaging. It will be administered intravenously on the day of imaging. Subjects will receive a bolus injection of 9mCi (331 MBq) of [18F]DCFPyL through a peripheral IV catheter. 60 to 120 minutes after injection, a whole body (toes to vertex) lowdose CT will be obtained (120 kVp, 80 mA maximum).
  Other Names: [18F]DCFPyL (PyL)
Procedure: PET/CT imaging — As per standard of care, acquisition will be performed on PET/CT scanner (Siemens, Germany) operating in 3D emission mode with CT-derived attenuation correction.
  Other Names: PET/CT acquisition

SUMMARY:
Primary Objective:

* To determine whether changes in uptake of [18F]DCFPyL PET/CT scans at baseline and after 6 weeks of treatment for metastatic castrate resistant prostate cancer, correlates with radiographic progression free survival (rPFS) as defined by Prostate Cancer Working Group 3 (PCWG3) criteria.

Secondary Objectives:

* To determine whether changes in uptake of [18F]DCFPyL PET/CT scans correlate with overall survival (OS)
* To determine whether baseline SUVmax correlate with rPFS
* To compare number of lesions detected with standard imaging at baseline and at the time of progression

DETAILED DESCRIPTION:
Prostate cancer is the most common cancer and the third most common cause of cancer deaths in American men. The lethal form of the disease is metastatic castrate resistant prostate cancer (mCRPC). Serum prostate specific antigen (PSA) testing has been relied upon heavily as a marker of disease and is commonly used in the community to guide therapy.

PyL, also known as [18F]DCFPyL, is a second-generation fluorinated prostate-specific membrane antigen (PSMA) targeted positron emission tomography (PET) imaging agent. In preliminary studies it demonstrates a higher detection of metastatic prostate lesions compared to standard imaging. However, the role of [18F] PyL in tumor response to therapy has not been evaluated, specifically the potential to serve as a predictive biomarker of response. Given the high cost of current therapeutic agents in mCRPC, there is a need for an early response biomarker to stratify which patients will benefit from therapy and which will not. This will also allow for earlier change in management of patients who will not response to these therapies, potentially improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of prostate cancer
* Age ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Metastatic castrate resistant prostate cancer as defined by Prostate Cancer Working Group 3
* Eligible to receive systemic treatment (abiraterone, enzalutamide, docetaxel, cabazitaxel) for their disease
* Ability to understand and willingness to sign a written informed consent document
* Wiling to comply with clinical trial instructions and requirements

Exclusion Criteria:

* History of another active malignancy within 3 years, other than basal cell and squamous cell carcinoma of the skin
* Presence of prostate brachytherapy implants
* Administration of another radioisotope within five physical half-lives of trial enrollment
* Radiation or chemotherapy within 2 weeks prior to trial enrollment
* Serum creatinine > 3 times the upper limit of normal
* Serum total bilirubin > 3 times the upper limit of normal
* Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) >5 times the upper limit of normal
* Inadequate venous access

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of changes in PyL PET imaging correlating with radiographic Progression-Free Survival (rPFS) | Baseline, Post-treatment (approximately 6 weeks)
  To determine if changes in PyL PET/CT scans before and after 6 weeks on treatment is associated with stability of disease as measured by standard imaging.

SECONDARY OUTCOMES:
Prevalence of changes in uptake of [18F]DCFPyL PET/CT scans correlating with Overall Survival (OS) | Baseline, Post-treatment (approximately 6 weeks)
  The percent difference in summed SUV between the first and second PET/CT will be noted.
Prevalence of baseline SUVmax correlating with rPFS | Baseline, Post-treatment (approximately 6 weeks)
  To determine if standardized uptake values (SUVs) at baseline is a good measure for patient evaluation.
Change in number of lesions detected with standard imaging at baseline and at the time of progression | Baseline, up to 1 year
  To compare lesions detected with standard imaging

CONTACTS AND LOCATIONS:
Overall Officials: Matthew C. Dallos, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer Statistics, 2017. CA Cancer J Clin. 2017 Jan;67(1):7-30. doi: 10.3322/caac.21387. Epub 2017 Jan 5. PMID 28055103
- [Background] Szabo Z, Mena E, Rowe SP, Plyku D, Nidal R, Eisenberger MA, Antonarakis ES, Fan H, Dannals RF, Chen Y, Mease RC, Vranesic M, Bhatnagar A, Sgouros G, Cho SY, Pomper MG. Initial Evaluation of [(18)F]DCFPyL for Prostate-Specific Membrane Antigen (PSMA)-Targeted PET Imaging of Prostate Cancer. Mol Imaging Biol. 2015 Aug;17(4):565-74. doi: 10.1007/s11307-015-0850-8. PMID 25896814
- [Background] Rowe SP, Macura KJ, Mena E, Blackford AL, Nadal R, Antonarakis ES, Eisenberger M, Carducci M, Fan H, Dannals RF, Chen Y, Mease RC, Szabo Z, Pomper MG, Cho SY. PSMA-Based [(18)F]DCFPyL PET/CT Is Superior to Conventional Imaging for Lesion Detection in Patients with Metastatic Prostate Cancer. Mol Imaging Biol. 2016 Jun;18(3):411-9. doi: 10.1007/s11307-016-0957-6. PMID 27080322